CLINICAL TRIAL: NCT01464541
Title: Orbital Fractures Measurement: Intraoperative Versus Computed Tomography (CT) Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EMC-0046-11
Record Dates: First submitted 2011-10-18; First posted 2011-11-03 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Orbital Fractures
Keywords: Orbit; Fracture; measurement; CT; intraoperative
MeSH Terms: conditions — Orbital Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- orbital fractures size (Experimental): patients who undergo surgical repair of orbital fracture with measuring the fracture size intraoperatively and had available orbital Ct scan preoperatively.
  Interventions: Procedure: operative fracture size vs CT fracture size; Procedure: orbital fracture intraoperative measurement

INTERVENTIONS:
Procedure: operative fracture size vs CT fracture size — comparing actual intraoperative fracture size to the CT fracture size
Procedure: orbital fracture intraoperative measurement — comparing intraoperative fracture size to the CT orbital fracture size

SUMMARY:
Purpose to compare the orbital fracture size measured by orbital CT scan and compare it to the actual orbital fracture size intraoperatively in patients who needed surgical intervention to correct the fracture.

Hypothesis: there is difference between the CT measure fracture size and the actual intraoperative size.

ELIGIBILITY:
Inclusion Criteria:

* With orbital fracture (trauma) proved by CT scan and need operative repair.
* Agree to participate.

Exclusion Criteria:

* Patients that refuse to be included in the study.
* Under the age of 18 years.
* CT not performed or not available.
* Not qualified to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Patients with orbital fractures that require surgical repair will have their fracture"s" size measured intraoperatively by a ruler and/or a caliper in millimeters and compare it to the size measured by the CT scan. | 2 years
  Patients with orbital fractures that need to be operated. Their intraoperative fracture size will be measured by the orbital surgeon by a ruler or/and a caliper in millimeters. Size on CT scan is determined by counting the number of slides that show the fracture (for anteropsterior fracture we measure the number of coronal sections that show the fracture multiply X1-each section is 1millimeter thickness, and so on for mediolateral fractures we measure saggital sections number and for superoinferior fractures the axial sections that show the fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Briscoe, MD, Principal Investigator — Chairperson, dept. of ophthalmology, haemek medical center, afula 18101, Israel; Wasseem Hilo, MD, Study Director — Resident, ophthalmology dept, Haemek Medical Center, Afula 18101, Israel
Locations (2):
- Israel (2):
  - HaEmek medical center, Afula, North
  - HaEme Medical center, Dept of Ophthalmology, Afula